CLINICAL TRIAL: NCT01138163
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial of Bavituximab Plus Docetaxel in Patients With Previously Treated Locally Advanced or Metastatic Non-Squamous Non Small-Cell Lung Cancer
Brief Title: Study of Bavituximab Plus Docetaxel in Patients With Locally Advanced or Metastatic Non-Squamous Non Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPHM 0902
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Non-small-cell Lung Cancer
Keywords: NSCLC; second-line; lung cancer; non small cell lung cancer; bavituximab; monoclonal antibody
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel; bavituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Docetaxel plus bavituximab 1 mg/kg (Experimental)
  Interventions: Drug: Docetaxel plus bavituximab or placebo
- Docetaxel plus bavituximab 3 mg/kg (Experimental)
  Interventions: Drug: Docetaxel plus bavituximab or placebo
- Docetaxel plus placebo (Placebo Comparator)
  Interventions: Drug: Docetaxel plus bavituximab or placebo

INTERVENTIONS:
Drug: Docetaxel plus bavituximab or placebo — Patients will be randomized to receive docetaxel plus placebo, docetaxel plus 1 mg/kg bavituximab, or docetaxel plus 3 mg/kg bavituximab in the Combination Therapy Period. The Combination Treatment Period for each patient will begin on Study Day 1. Docetaxel, 75 mg/m2, will be given on Day 1 of each 21 day cycle for up to 6 cycles, and placebo or the assigned dose of bavituximab will be given weekly. Docetaxel administration will occur every 21 days. All patients who complete the Combination Therapy Period (or discontinue for any reason other than disease progression or toxicity) will be eligible to enter the Monotherapy Period. Patients will continue to receive assigned blinded treatment (placebo or 1 or 3 mg/kg bavituximab) weekly until progression or toxicity.

SUMMARY:
The primary purpose of this research study is to see whether adding bavituximab (an investigational drug) to the standard chemotherapy drug docetaxel, will improve the results of the treatment for non-small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18 years of age with a life expectancy of at least 3 months.
* Histologically or cytologically confirmed stage IIIB or stage IV non squamous non-small-cell lung cancer (NSCLC) who have progressed after 1 chemotherapy regimen.
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST, Version 1.1) on cross-sectional imaging that is at least 2 cm in longest diameter.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Adequate hematologic, renal, and hepatic function.
* PT/INR ≤ 1.5 × ULN; aPTT time ≤ 1.5 × ULN.
* New York Heart Association classification I or II

Exclusion Criteria:

* Squamous, small cell, or mixed histology.
* Known history of bleeding diathesis or coagulopathy.
* Cavitary tumors or tumors invading or abutting large blood vessels.
* Bleeding: Clinically significant bleeding such as gross hematuria, GI bleeding and hemoptysis within 12 months of Screening.
* Venous thromboembolic events within 6 months of screening.
* Ongoing therapy with oral or parenteral anticoagulants.
* Concurrent estrogens, anti-estrogens or progesterone compounds.
* Radiotherapy within 2 weeks or major surgery within 4 weeks preceding Study Day 1.
* Symptomatic or clinically active brain metastases.
* Symptomatic coronary artery disease, cerebrovascular accident, transient ischemic attack, myocardial infarction or unstable angina pectoris within 6 months of screening.
* Grade 2 or higher peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Until disease progression

CONTACTS AND LOCATIONS:
Locations (53):
- United States (24):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - South Bay Hematology Oncology, Campbell, California
  - Medical Oncology Care Associates, Orange, California
  - American Institute of Research, Whittier, California
  - The Center for Hematology-Oncology/Boca Raton Community Hospital, Inc, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Georgia Cancer Specialists, PC, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Cedar Valley Medical Specialists, PC, Waterloo, Iowa
  - Jewish Hospital, Louisville, Kentucky
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Nebraska Hematology Oncology, PC, Lincoln, Nebraska
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - The Christ Hospital Cancer Center Research, Cincinnati, Ohio
  - Oncology/ Hematology Care, Inc, Cincinnati, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Pennsylvania State Hershey Cancer Institute, Hershey, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Hospitals and Clinics, Huntsman Cancer Institute, Salt Lake City, Utah
- Georgia (2):
  - JSC A.Gvamichava National Oncology Center, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
- India (15):
  - BiBi General Hospital & Cancer Centre, Hyderabad, Andhra Pradesh
  - Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Mahavir Cancer Sansthan, Patna, Bihar
  - O.P. Jindal Institute of Cancer & Research, Hisar, Haryana
  - Bangalore Institute of Oncology Specialty Centre, Bangalore, Karnataka
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - Bharath Hospital and Institute of Oncology, Mysore, Karnataka
  - Kodlikeri Memorial Hospital, Aurangabad, Maharashtra
  - Cancer Care Clinic, Nagpur, Maharashtra
  - Shatabdi Superspecialty Hospital, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - SMS Medical College Hospital, Jaipur, Rajasthan
  - Chhatrapati Shahuji Maharaj Medical University, Lucknow, Uttar Pradesh
  - Shanti Mukund Hospital Curie Cancer Center, Delhi
  - All India Institute of Medical Sciences, Delhi
- Russia (7):
  - State Medical Preventive Institution "Chelyabinsk Regional Clinical Oncology", Chelyabinsk
  - State Institution of Healthcare " Ivanovo Regional Oncology Dispensary ", Ivanovo
  - Institution of Russian Academy of Medical Science "Russian Oncology Scientific Centre named after N. N. Blokhina RAMN", Moscow
  - State Educational Institution of Higher Professional Education "Saint-Petersburg State Medical University named after academician I.P. Pavlov of Federal Agency of Healthcare and Social Development", Saint Petersburg
  - State Institution of Healthcare "Pyatigorsk Oncology Dispensary", Stavropol
  - State Institution of Healthcare "Tula Regional Oncology Dispensary", Tula
  - State Institution of Healthcare of Yaroslavl Region "Regional Clinical Oncology Hospital", Yaroslavl
- Ukraine (5):
  - City multi-field clinical hospital # 4, Department of chemotherapy; Dnipropetrovsk State Medical Academy, Chair of Oncology and Medical Radiology;, Dnipropetrovsk
  - Municipal Clinical Medical and Prophylactic Institution "Donetsk Regional Antineoplastic Center", onco-chemotherapy, Donetsk
  - State Institution "Institute of Medical Radiology named after S.P. Grygoryev of AMS of Ukraine", department of chemotherapy, Kharkiv
  - Kyiv City Oncology Hospital, Thoracal Department, Kyiv
  - Uzhgorod Central City Clinical Hospital, City Oncology Center, Uzhhorod